CLINICAL TRIAL: NCT06909578
Title: Microvascular Obstruction Diagnosis Using the CoFI™ System Assessment - II
Acronym: MOCA II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CorFlow Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2402
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Microvascular Obstruction (MVO); STEMI - ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Adult subjects presenting with STEMI in the LAD undergoing PPCI (Other)
  Interventions: Device: CorFlow Controlled Flow Infusion System - CoFI™

INTERVENTIONS:
Device: CorFlow Controlled Flow Infusion System - CoFI™ — The CorFlow CoFI™ System is intended to assess the dynamic microvascular resistance and to treat microvascular obstruction in the coronary vasculature of patients following PCI with stent placement.

SUMMARY:
A prospective, multicenter, international single-arm, pivotal clinical study designed to validate the performance of the CoFI system in detecting MVO in STEMI subjects, as confirmed by CMRI. The study will be conducted in accordance with the Declaration of Helsinki, EN ISO 14155:2020, local and national regulations.

Each study site will receive support from a sponsor-certified proctor during the learning curve to ensure consistent and accurate application of the CoFI system.

DETAILED DESCRIPTION:
Microvascular obstruction (MVO) is a common complication that occurs after establishing coronary vessel patency by percutaneous coronary intervention (PCI) for the treatment of acute myocardial infarction (AMI).

Despite the successful restoration of vessel patency through PCI, 50% to 70% of STEMI subjects experience MVO, which affects vessels in the myocardial microcirculation. MVO occurs most commonly in the setting of AMI because the prolonged ischemia leads to endothelial damage, myocyte oedema and microvascular dysfunction.

Research has shown that MVO increases the risk of poor clinical outcomes, including death, re-infarction, reduced left ventricular ejection fraction (LVEF), left ventricular (LV) remodeling, heart failure, and more.

Late gadolinium enhancement (LGE) cardiac magnetic resonance imaging (CMRI) is the current state-of-the-art for MVO identification and quantification. However, due to clinical reasons, CMRI imaging cannot be performed during the subject's emergent state. In most cases, this means that the diagnosis is made outside the biological window where MVO-related damage to heart muscle could be reversed or at least reduced.

Thus, although CMRI is the most accurate method to diagnose MVO, its use in routine practice is limited. Therefore, a direct and accurate quantitative diagnosis during primary PCI is required for early risk stratification in routine clinical practice.

The Controlled Flow Infusion (CoFI) system is designed to be integrated into current PCI protocols, enabling the rapid and safe detection of MVO after successful PCI procedures. Using a proprietary algorithm, the system can provide an output for diagnosing microvascular obstruction (MVO) immediately post-PCI by measuring real-time distal coronary back-pressure response to a dynamic infusion sequence downstream of a low-pressure occlusion balloon.

The aim of the study is to validate the diagnostic performance of the CoFI system in detecting MVO in anterior STEMI subjects following PPCI as measured in CMRI 1-3 days post-procedure.

The study has two phases 1 & 2. Phase 1 aims to demonstrate whether the pCoFI threshold for MVO detection gathered in the US population aligns with the 95% confidence interval (CI) of the pCoFI threshold from the EU population gathered in the FIH MOCA-I study. Phase 2 has two possible routes, A or B. Depending on the outcome of phase 1, the study will continue along either route. The study progresses into pivotal route A if the threshold 95% CI aligns as described above and into route B if it does not. If the study follows route B the threshold will be reset and the sample size recalculated. In case of route B phase 1 data will become part of the data training set, whereas in route A would phase 1 data will be included in the study analysis set.

With a need to follow Route B, comes a substantial clinical investigation plan (CIP) amendment/supplement submission to the FDA and applicable IRBs, before restarting the study.

The sample size for the MOCA-II feasibility and pivotal phases will be based on a conservative assumed disease prevalence of 50% MVO+.

Interim Analysis An interim analysis is planned to be done after 50% of the subjects have been enrolled to verify if the study's success or futility criteria are met.

Based on the interim analysis, the sample size for the primary endpoint may be adjusted according to the actual MVO prevalence from the study data set, as defined by CMRI at 1 to 3 days post-PPCI. The observed prevalence and interim estimates of sensitivity and specificity will be used to reassess the required sample size if the interim study data do not justify an early stop for success.

ELIGIBILITY:
Inclusion Criteria:

* Clinical:

  1. Subject ≥18 years of age
  2. Ability to provide written informed consent according to GCP and governing regulations
  3. Diagnosis of acute anterior STEMI
  4. Persistent symptoms to balloon time ≤ 6 hours. The assessment by the treating investigator after evaluation by subjects explanation is the defining timepoint for symptom onset.

PPCI & Angiographic

1. Culprit lesion in the LAD
2. COFI ballon can be placed according to IFU
3. Required stent diameter ≥ 2.75 mm and ≤ 5mm
4. Required stent length ≥ 15 mm
5. Successful PPCI Procedure as documented by <50% diameter residual angiographic stenosis within all treated culprit lesions with TIMI 2 or 3 flow.

Exclusion Criteria:

* Clinical:

  1. Cardiogenic shock
  2. Thrombolytic therapy administered for this STEMI
  3. Contraindication to CMRI

     1. Cardiac pacemaker or implantable defibrillator;
     2. Non-MRI compatible aneurysm clip;
     3. Neural Stimulator (i.e., TENS unit);
     4. Any implanted or magnetically activated device (insulin pump);
     5. Any type of non-MRI compatible ear implant;
     6. Metal shavings in the orbits;
     7. Any metallic foreign body, shrapnel, or bullet in a location which the physician feels would present a risk to the subject;
     8. Any history indicating contraindication to MRI
     9. Inability to follow breath hold instructions or to maintain a breath hold for >15 seconds; and
     10. Known hypersensitivity or contraindication to gadolinium contrast.
  4. Subject with previous MI and/or known cardiomyopathy (ischemic and non ischemic), ventricular pseudoaneurysm, VSD, severe mitral valve regurgitation (with or without papillary muscle rupture), severe known cardiac valvular stenosis or insufficiency, pericardial disease
  5. Major bleeding ≤ 30d prior to intervention
  6. Major surgery ≤ 30d prior to intervention
  7. TIA or stroke ≤ 30d prior to intervention
  8. Heart failure with inotrope support and/or consideration for LVAD or heart transplant
  9. Known severe renal disease with creatinine > 2.5 mg/dL and/or eGFR < 30 mL/min/1.73 m2
  10. Subject has other medical illness (e.g., cancer, dementia) or known history of substance abuse (alcohol, cocaine, heroin, etc.) that may cause non-compliance with the CIP, confound the data interpretation, or is associated with limited life expectancy of less than one year
  11. Current participation in another clinical study
  12. Pregnancy

PPCI & Angiographic:

1. CABG of LAD
2. Unsuitable target vessel anatomy (excessive tortuosity, diffuse disease, or moderate/heavy calcification)
3. Cardiac condition preventing the use of the CoFI System
4. Any angiographic post stenting condition that according to the physician implies soc administration of any GpIIb/IIIa inhibitors or adenosine
5. Cardiac condition mandating elective PCI/CABG procedure prior to CMRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | From enrollment to the end of treatment at 6 Months
  Diagnostic performance is measured by sensitivity and specificity of the CoFI system in detecting MVO in relation to the pre-set PCoFI threshold of 124 mmHg. The analysis will be per-protocol (PP) (primary) and the full analysis set (FAS) (secondary).
  Hypothesis
  Sensitivity and Specificity will be tested to meet the acceptance criteria:
  i.The lower bound of the confidence interval (CI) for sensitivity is 70% ii. The lower bound of the CI for specificity is 65% H0: p < p0 H1: p ≥ p0 p0 = 70%se, 65%sp

IPD SHARING:
Plan to Share IPD: No
Decide has to made by study leadership.